CLINICAL TRIAL: NCT04724590
Title: OPHTHALMOLOGIC EVALUATION OF RADIATION-RELATED OPTIC NEUROPATHY FOLLOWING IMAGE GUIDED INTENSITY-MODULATED RADIATION THERAPY (IMRT) FOR NASOPHARYNGEAL CARCİNOMA (ORONIN)
Brief Title: OPHTHALMOLOGIC EVALUATION OF RADIATION-RELATED OPTIC NEUROPATHY FOLLOWING IMAGE GUIDED INTENSITY-MODULATED RADIATION THERAPY (IMRT) FOR NASOPHARYNGEAL CARCİNOMA
Acronym: ORONIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Meltem Dağdelen, MD, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 83045809-604.01.02; 159075 (Other: IstanbulUC)
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: The Aim of Our Study is to Prospectively Evaluate the Optic Neuropathy in Nasopharynx Cancer Patients
Keywords: RADIATION-RELATED OPTIC NEUROPATHY,NASOPHARYNGEAL CARCİNOMA, RADIOTHERAPY
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: IMRT(IMAGE GUIDED INTENSITY-MODULATED RADIATION THERAPY ) — Evaluation the optic neuropathy in nasopharynx cancer patients treated in our clinic.
  Other Names: OCT(Optical Coherence Tomography), OCT-A(Optical Coherence Tomography Angiography)

SUMMARY:
Primary treatment in nasopharynx cancers is radiotherapy (RT) or chemoradiotherapy (CRT) depending on the stage of the tumor. According to the guidelines, the dose of radiotherapy for primary tumors varies between 66-70 Gy. In consideration of modern radiotherapy techniques like IMRT with systemic chemotherapy for nasopharyngeal cancer, loco-regional control has been perfect. However, the rate of late complications from treatment, many of which are irreversible, is still high. Radiation-related optic neuropathy is the late complication that optic nerves might be affected during the radiotherapy due to the close location of the nasopharynx. Incidence of this is 8.7-9% in head and neck cancer and is observed between 2-9 years after RT. Painless, irreversible, and progressive vision loss usually occurs, and the pallor of optic disc margins, retinal vein dilatation, bleeding, and neovascularization are in the ophthalmic examination. The risk of optic neuropathy increases when the tumor is in close contact with optic nerves, radiation dose, concurrent chemotherapy used, history of diabetes or hypertension.

The aim of our study is to prospectively evaluate optic neuropathy in nasopharynx cancer patients treated in our clinic.

ELIGIBILITY:
Inclusion Criteria:

Patient with nasopharyngeal carcinoma that histopathologically confirmed Age >18 Radiotherapy or chemoradiotherapy applied to the patient in our clinic No recurrence or metastasis during follow-up Optic evaluation Evaluation with MRI or CT during follow-up

Exclusion Criteria:

Cranial RT No histopathological verification Age< 18 There were locoregional recurrence or metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-04-03 (Estimated); Study Completion 2021-05-03 (Estimated)

PRIMARY OUTCOMES:
OPHTHALMOLOGIC EVALUATION OF RADIATION-RELATED OPTIC NEUROPATHY FOLLOWING IMAGE GUIDED INTENSITY-MODULATED RADIATION THERAPY (IMRT) FOR NASOPHARYNGEAL CARCİNOMA (ORONIN) RADIATION-RELATED OPTIC NEUROPATHY | 2-9 years
  RADIATION-RELATED OPTIC NEUROPATHY

CONTACTS AND LOCATIONS:
Locations (1):
- Meltem Dağdelen, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided